CLINICAL TRIAL: NCT00967616
Title: Randomized, Active-Controlled, Open-Label Phase 2 Study of CS-7017 in Combination With FOLFIRI in Subjects With Metastatic Colorectal Cancer Who Failed First-Line Therapy
Brief Title: Study of CS-7017 in Combination With FOLFIRI in Subjects With Metastatic Colorectal Cancer Who Failed First-Line Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CS7017-A-U203
Record Dates: First submitted 2009-08-27; First posted 2009-08-28 (Estimated); Results first posted 2020-05-04 (Actual); Last update posted 2020-05-04 (Actual); Status verified 2020-04

CONDITIONS: Colorectal Cancer; Neoplasms, Colorectal
Keywords: metastatic; colon; rectum; combination; chemotherapy
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — efatutazone; Irinotecan; Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- FOLFIRI (Active Comparator): Participants who received irinotecan, leucovorin, and 5-fluorouracil (5-FU) (FOLFIRI). FOLFIRI was administered by intravenous (IV) injection once every 2 weeks. The FOLFIRI regimen consisted of:
  * Irinotecan, 180 mg/m^2 IV infusion over 30 to 120 minutes
  * Leucovorin, 400 mg/m^2 IV infusion to match the duration of the irinotecan infusion
  * 5-FU, 1200 mg/m^2/day x 2 days (total 2400 mg/m^2 over 46 to 48 hours continuous infusion)
  Interventions: Drug: irinotecan, leucovorin, and 5-fluorouracil (5-FU) (FOLFIRI)
- CS7017+FOLFIRI (Experimental): Participants who received CS7017 plus irinotecan, leucovorin, and 5-fluorouracil (5-FU) (FOLFIRI). Two CS-7017 tablets were administered by mouth (PO) twice a day (BID) every 12 hours. FOLFIRI was administered IV once every 2 weeks. The FOLFIRI regimen consisted of:
  * Irinotecan, 180 mg/m^2 IV infusion over 30 to 120 minutes
  * Leucovorin, 400 mg/m^2 IV infusion to match the duration of the irinotecan infusion
  * 5-FU, 1200 mg/m^2/day x 2 days (total 2400 mg/m^2 over 46 to 48 hours continuous infusion)
  Interventions: Drug: CS7017; Drug: irinotecan, leucovorin, and 5-fluorouracil (5-FU) (FOLFIRI)

INTERVENTIONS:
Drug: CS7017 — CS-7017 (0.25mg tablet) Two CS-7017 tablets will be administered by mouth (PO) BID every 12 hours. FOLFIRI will be administered IV once every 2 weeks.
  Arms: CS7017+FOLFIRI
Drug: irinotecan, leucovorin, and 5-fluorouracil (5-FU) (FOLFIRI) — FOLFIRI will be administered IV once every 2 weeks.
  The FOLFIRI regimen consists of:
  * Irinotecan, 180 mg/m^2 IV infusion over 30 to 120 minutes
  * Leucovorin, 400 mg/m^2 IV infusion to match the duration of the irinotecan infusion
  * 5-FU, 1200 mg/m^2/day x 2 days (total 2400 mg/m^2 over 46 to 48 hours continuous infusion)
  Other Names: Irinotecan; Leucovorin; 5-FU; 5-fluorouracil

SUMMARY:
This phase 2, randomized, active-controlled, open-label, parallel group, multicenter study will be conducted at up to 18 study centers in the US, Central America, and South America. Adult subjects with metastatic colorectal cancer (CRC) who failed first-line chemotherapy will participate in the study, which will be conducted on an outpatient basis. It is anticipated that 100 subjects will be enrolled to obtain approximately 90 evaluable subjects.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic CRC that has progressed following first-line therapy.
* Measurable disease (Response Evaluation Criteria in Solid Tumors [RECIST], Version 1.0.
* Male or female ≥ 18 years of age.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
* Resolution of any toxic effects of prior therapy (except alopecia) to NCI CTCAE, Version 3.0, grade ≤ 1.
* Adequate organ and bone marrow function as evidenced by:

  * Hemoglobin ≥ 9 g/dL (transfusion and/or growth factor support allowed)
  * Absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L
  * Platelet count ≥ 100 x 10^9/L
  * Serum creatinine ≤ 1.5 x the upper limit of normal (ULN) or creatinine clearance ≥ 60 mL/min
  * Aspartate aminotransferase (AST) and alkaline phosphatase ≤ 2.5 x ULN in participants with no liver metastasis and ≤ 5.0 x ULN in participants with liver metastasis
  * Total bilirubin ≤ 1.5 x ULN
* Women of childbearing potential must be willing to consent to using effective contraception (eg, hormonal contraceptives, bilateral tubal ligation, barrier with spermicide, intrauterine device) while on treatment and for at least 3 months thereafter. Men who are the partner of a woman of childbearing potential must be willing to consent to using effective contraception (eg, vasectomy or barrier with spermicide) while on treatment and for 3 months thereafter.
* All female participants of childbearing potential must have a negative pregnancy test (serum or urine) result before initiating study treatment.
* Participants must be fully informed about their illness and the investigational nature of the study protocol (including foreseeable risks and possible side effects) and must sign and date an Independent Ethics Committee (IEC)- or Institutional Review Board (IRB)-approved informed consent form (ICF) (including HIPAA authorization, if applicable) before performance of any study-specific procedures or tests.
* Participants must be willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* First-line treatment with an irinotecan-based regimen (eg, FOLFIRI).
* Anticipation of need for a major surgical procedure or radiation therapy (RT) during the study.
* Treatment with chemotherapy, other thiazolidinediones (TZD), RT, surgery, immunotherapy, biological therapy, or any investigational anticancer agent within 4 weeks before start of study treatment.
* History of any of the following conditions within 6 months before initiating study treatment:

  * Diabetes mellitus requiring treatment with insulin or TZD agents
  * Myocardial infarction with significant impairment of cardiac function (eg, ejection fraction ≤ 50%)
  * Severe/unstable angina pectoris
  * Coronary/peripheral artery bypass graft
  * New York Heart Association (NYHA) class III or IV congestive heart failure
  * Malabsorption syndrome, chronic diarrhea (lasting > 4 weeks), inflammatory bowel disease, or partial bowel obstruction.
* Participants with clinically active brain metastases (defined as untreated, symptomatic, or requiring therapy with steroids or anticonvulsants to control associated symptoms); uncontrolled seizure disorder; spinal cord compression; or carcinomatous meningitis. Participants with treated brain metastasis will be included in the study if they have recovered from the acute, toxic effects of RT. A minimum of 15 days must have elapsed between the end of RT and enrollment into the study.
* History of malignancy other than CRC, unless there is an expectation that the malignancy has been cured, and tumor-specific treatment for the malignancy has not been administered within the previous 5 years.
* Clinically significant, severe, active infection requiring IV antibiotic or antiviral agents.
* Pericardial or pleural effusion (eg, requiring drainage) or pericardial involvement with the tumor. Participants with minimal pleural effusion may be eligible upon request by Investigator and approval by Sponsor.
* Need for concomitant use of other TZD agents during the study.
* Previous administration of CS-7017.
* Pregnant or breast feeding.
* Known to be homozygous for the UGT1A1*28 allele.
* Known history of severe hypersensitivity reactions to any of the components of CS-7017, irinotecan, leucovorin, or 5-FU.
* Serious intercurrent medical or psychiatric illnesses or any other conditions that in the opinion of the Investigator would impair the ability to give informed consent or unacceptably reduce protocol compliance or safety of the study treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-09; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (17):
- United States (6):
  - Beverly Hills Cancer Center, Beverly Hills, California
  - St. Jude Heritage Medical Group, Fullerton, California
  - John Marshall, Washington D.C., District of Columbia
  - Georgia Cancer Specialists, Atlanta, Georgia
  - Victor Priego, Bethesda, Maryland
  - Gabrail Cancer Center, Canton, Ohio
- Argentina (2):
  - Instituto FIDES Oncologia y Especialidades Medicas, Buenos Aires
  - CAIPO Centro para la Atencion Integral del Paciente Oncologico, San Miguel de Tucumán
- Brazil (3):
  - Hospital Sao Lucas da Pontificia Universidade Catolica do Rio Grande do Sul - PUC-RS, Porto Alegre
  - Instituto Nacional de Cancer INCA, Rio de Janeiro
  - ICAVC, São Paulo
- Chile (3):
  - Fundacion Arturo Lopez Perez, Santiago
  - Instituto Nacional del Cancer, Santiago
  - Instituto Oncologico Clinica Renaca, Viña del Mar
- Peru (3):
  - Hospital Nacional Alberto Sabogai Sologuren, Callao
  - Hospital Nacional Dos de Mayo, Lima
  - Oncosalud SAC, Lima

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 100 participants who met all inclusion and no exclusion criteria were randomized to treatment in the study.
Groups:
- CS7017 + FOLFIRI: Participants who received CS7017 plus irinotecan, leucovorin, and 5-fluorouracil (5-FU) (FOLFIRI). Two CS-7017 tablets were administered PO BID every 12 hours. FOLFIRI was administered IV once every 2 weeks. The FOLFIRI regimen consisted of:
  * Irinotecan, 180 mg/m^2 IV infusion over 30 to 120 minutes
  * Leucovorin, 400 mg/m^2 IV infusion to match the duration of the irinotecan infusion
  * 5-FU, 1200 mg/m^2/day x 2 days (total 2400 mg/m^2 over 46 to 48 hours continuous infusion)
Period: Overall Study
Arm/Group | FOLFIRI | CS7017 + FOLFIRI
Started | 50 | 50
Completed | 0 | 0
Not Completed | 50 | 50
Not completed — Adverse Event or Serious Adverse Event | 2 | 17
Not completed — Death | 0 | 3
Not completed — Withdrawal by Subject | 8 | 4
Not completed — Progressive Disease | 31 | 18
Not completed — Other | 8 | 8
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FOLFIRI | CS7017 + FOLFIRI | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 31 | 64
  >=65 years | 17 | 19 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (12.36) | 59.7 (11.79) | 59.0 (12.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 22 | 44
  Male | 28 | 28 | 56
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 4 | 11
  White | 42 | 38 | 80
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 6 | 7

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Progression-Free Survival at 16 Weeks After Administration of CS-7017 Combined With Irinotecan, Leucovorin, and 5-Fluorouracil (5-FU) After Failure of First-line Therapy in Treatment of Metastatic Colorectal Cancer
Description: Progression-free survival (PFS) was defined as the time from randomization until the first objective evidence of disease progression or death from any cause.
Time Frame: Baseline to 16 weeks postdose
Population: PFS was assessed in the Full Analysis Set.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | FOLFIRI | CS7017 + FOLFIRI
Number analyzed (Participants) | 50 | 50
percentage of participants | 66.7 [53.6 to 76.9] | 59.7 [45.6 to 71.2]

2. Secondary Outcome: Median Overall Progression-Free Survival Following Administration of CS-7017 in Combination With Irinotecan, Leucovorin, and 5-Fluorouracil (5-FU) (FOLFIRI) After Failure of First-line Therapy in Treatment of Metastatic Colorectal Cancer
Description: as for outcome 1
Time Frame: Baseline to approximately 3 years postdose
Population: PFS was assessed in the Full Analysis Set.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | FOLFIRI | CS7017 + FOLFIRI
Number analyzed (Participants) | 50 | 50
months | 4.2 [3.8 to 5.6] | 4.4 [3.5 to 7.2]

3. Secondary Outcome: Median Overall Progression-Free Survival: Sensitivity Analysis Including Clinical Progression After Administration of CS-7017 and Irinotecan, Leucovorin, and 5-Fluorouracil After Failure of First-line Therapy of Metastatic Colorectal Cancer
Description: Progression-free survival (PFS) was defined as the time from randomization to the date of the first objective documentation of progressive disease (PD) or death resulting from any cause, whichever came first. The sensitivity analysis included clinical progression as an event.
Time Frame: Baseline to approximately 3 years postdose
Population: PFS was assessed in the Full Analysis Set.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | FOLFIRI | CS7017 + FOLFIRI
Number analyzed (Participants) | 50 | 50
months | 4.2 [3.7 to 5.6] | 4.4 [3.5 to 7.2]

4. Secondary Outcome: Best Overall Response and Objective Response Rate Following Administration of CS-7017 in Combination With Irinotecan, Leucovorin, and 5-Fluorouracil (FOLFIRI) After Failure of First-line Therapy in Treatment of Metastatic Colorectal Cancer
Description: As per Response Evaluation Criteria for Solid Tumors v1.0, best overall response was characterized as confirmed complete response (CR) defined as disappearance of all target lesions, confirmed partial response (PR) defined as ≥30% decrease from baseline, stable disease (SD) defined as neither progressive disease (PD) nor PR, and PD defined as ≥20% increase from smallest sum of longest diameter recorded since treatment started. Objective response rate (ORR) was defined as CR + PR. If there is no tumor assessment after the first dose of study drug, the best overall response is classified as Inevaluable.
Time Frame: Baseline to approximately 3 years postdose
Population: Best overall response and response rates were assessed in the Full Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | FOLFIRI | CS7017 + FOLFIRI
Number analyzed (Participants) | 50 | 50
Participants
  Confirmed CR | 0 | 0
  Confirmed PR | 7 | 10
  Objective response (confirmed CR+PR) | 7 | 10
  Stable disease | 29 | 18
  Progressive disease | 10 | 8
  Inevaluable | 2 | 12
  Best overall response of SD or better | 38 | 30

5. Secondary Outcome: Treatment-Emergent Adverse Events Occurring in ≥10% of Participants Following Administration of CS-7017 Combined With Irinotecan, Leucovorin, and 5-Fluorouracil (FOLFIRI) After Failure of First-line Therapy in Treatment of Metastatic Colorectal Cancer
Description: An adverse event (AE) >30 days after last dose of study drug was not included as a treatment-emergent adverse events (TEAE) unless considered related to treatment.
Time Frame: Baseline to 30 days post last dose, up to approximately 3 years
Population: Treatment-emergent adverse events were assessed in the Safety Analysis Set.
Measure: Count of Participants; unit: Participants
Arm/Group | FOLFIRI | CS7017 + FOLFIRI
Number analyzed (Participants) | 50 | 50
Participants
  Any TEAE | 50 | 50
  Blood and Lymphatic System Disorders | 24 | 42
  Anaemia | 16 | 35
  Febrile neutropenia | 0 | 7
  Leukopenia | 0 | 11
  Neutropenia | 10 | 33
  Thrombocytopenia | 2 | 9
  Eye Disorders | 1 | 8
  Gastrointestinal Disorders | 47 | 49
  Abdominal pain | 17 | 20
  Abdominal pain upper | 6 | 1
  Aphthous stomatitis | 5 | 2
  Constipation | 9 | 13
  Diarrhea | 33 | 30
  Nausea | 36 | 39
  Vomiting | 33 | 24
  General Disorders & Administration Site Conditions | 39 | 43
  Asthenia | 22 | 14
  Face Edema | 0 | 9
  Fatigue | 9 | 15
  Mucosal inflammation | 13 | 7
  Edema peripheral | 7 | 34
  Pyrexia | 5 | 10
  Infections & Infestations | 21 | 21
  Influenza | 5 | 1
  Injury, Poisoning, and Procedural Complications | 4 | 6
  Investigations | 16 | 28
  Weight decreased | 12 | 6
  Weight increased | 0 | 20
  Metabolism and Nutrition Disorders | 31 | 28
  Decreased appetite | 23 | 17
  Dehydration | 7 | 4
  Hypokalaemia | 4 | 6
  Musculoskeletal and Connective Tissue Disorders | 18 | 12
  Pain in extremity | 4 | 6
  Back pain | 6 | 3
  Nervous System Disorders | 17 | 14
  Dizziness | 5 | 3
  Headache | 3 | 5
  Psychiatric Disorders | 10 | 11
  Renal and Urinary Disorders | 6 | 9
  Reproductive System and Breast Disorders | 5 | 3
  Respiratory, Thoracic, and Mediastinal Disorders | 17 | 19
  Cough | 5 | 5
  Dyspnea | 7 | 6
  Skin and Subcutaneous Tissue Disorders | 21 | 20
  Alopecia | 11 | 10
  Vascular Disorders | 8 | 10

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse event data were collected from baseline to 30 days post last dose, up to approximately 3 years.
Description: Adverse events (AEs) were defined as any untoward, unfavorable, unintended medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. All-cause mortality includes all deaths that occurred during the study and within 30 days after the last dose of study drug.
Arm/Group | FOLFIRI | CS7017 + FOLFIRI
All-Cause Mortality (participants affected / at risk) | 2/50 | 7/50
Serious Adverse Events (participants affected / at risk) | 12/50 | 20/50
Other Adverse Events (participants affected / at risk) | 50/50 | 50/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FOLFIRI (N=50) | CS7017 + FOLFIRI (N=50)
Anaemia (Blood and lymphatic system disorders) | 3 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 6
Leukopenia (Blood and lymphatic system disorders) | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 2
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 0
Ascites (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Intestinal fistula (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 2
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 1 | 1
Asthenia (General disorders) | 1 | 1
Catheter site pain (General disorders) | 1 | 0
General physical health deterioration (General disorders) | 1 | 0
Generalised oedema (General disorders) | 0 | 1
Multi-organ failure (General disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 1
Jaundice (Hepatobiliary disorders) | 0 | 1
Device related infection (Infections and infestations) | 1 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 1
Endocarditis staphylococcal (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 0 | 1
Gastroenteritis Escherichia coli (Infections and infestations) | 0 | 1
Gingival infection (Infections and infestations) | 0 | 1
Neutropenic sepsis (Infections and infestations) | 0 | 1
Oral herpes (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Pulmonary sepsis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 2
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 1
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to bladder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to fallopian tube (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to ovary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to uterus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Haemorrhage urinary tract (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 2
Renal impairment (Renal and urinary disorders) | 0 | 1
Scrotal pain (Reproductive system and breast disorders) | 1 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Embolism venous (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | FOLFIRI (N=50) | CS7017 + FOLFIRI (N=50)
Anaemia (Blood and lymphatic system disorders) | 16 | 35
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 7
Leukopenia (Blood and lymphatic system disorders) | 0 | 11
Neutropenia (Blood and lymphatic system disorders) | 10 | 33
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 9
Abdominal pain (Gastrointestinal disorders) | 17 | 20
Diarrhea (Gastrointestinal disorders) | 33 | 30
Nausea (Gastrointestinal disorders) | 36 | 39
Vomiting (Gastrointestinal disorders) | 33 | 24
Asthenia (General disorders) | 22 | 14
Fatigue (General disorders) | 9 | 15
Edema peripheral (General disorders) | 7 | 34
Dehydration (Metabolism and nutrition disorders) | 7 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No